CLINICAL TRIAL: NCT05136963
Title: Development of a Bayesian Estimator for Calculating Plasma Iohexol Clearance Using Limited Sample Strategy for the Evaluation of Kidney Donation Candidates.
Brief Title: Development of a Bayesian Estimator for Calculating Plasma Iohexol Clearance
Acronym: CLIO
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19CH047; 2020-000853-29 (EudraCT Number)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Kidney Function Test
Keywords: iohexol; clearance; glomerular filtration flow rate; kidney donor
MeSH Terms: interventions — Iohexol; Pharmacokinetics; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteers (Experimental): 48 volunteers will be included according to the following demographic characteristics (corresponding to the demographic profile of kidney donors according to the national data of the Biomedicine Agency):
  * aged between 20 and 35 years old: 4 women, 3 men
  * aged between 35 and 50 years old: 7 women, 5 men
  * aged between 50 and 65: 11 women, 8 men
  * > 65 years old: 6 women, 4 men
  Interventions: Drug: Iohexol; Biological: pharmacokinetics

INTERVENTIONS:
Drug: Iohexol — 5 milliliter of iohexol will be administrated.
  Other Names: Omnipaque
Biological: pharmacokinetics — 10 blood samples of 5 milliliter will be performed. sampling time ater administration of Iohexol: 00h30, 1h00, 1h30, 02h00, 03h00, 04h00, 05h00, 06h00, 09h00 and 12h00
  Other Names: blood sample

SUMMARY:
In kidney transplantation, donor selection is based in part on the assessment of the functional capacity of the kidneys. For this purpose, it is recommended to measure the glomerular filtration rate (GFR) by a reference technique. To estimate GFR, several approaches are possible depending on the type of measurement (urinary or plasma) and the marker (exogenous or endogenous) used. Among these methods, the measurement of inulin clearance has long been considered the reference method. The occurrence of anaphylactic reactions led to its withdrawal from the market. Iohexol, an iodinated contrast agent, has characteristics similar to inulin. It is eliminated by glomerular filtration and its biological determination is simple.

Nevertheless, the techniques currently used to calculate plasma clearance of Iohexol have been imperfectly validated and are not always easy to implement in practice. the investigators propose to develop a Bayesian estimator for estimating Iohexol clearance applied to a population of healthy subjects, representative of potential kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated or entitled to a social security scheme
* Volunteers who has received informed information about the study and has co-signed, with the investigator, a consent to participate in the study.
* Aged > 18 years

Exclusion Criteria:

* Volunteers with a history or morbidities that would contraindicate assessment for kidney donation according to current recommendations
* Participation in another clinical research protocol within 3 months prior to inclusion
* Volunteers having hypersensitivity to Iohexol or one of its excipients
* Administration of iodinated contrast media in the week prior to inclusion
* Known history of an immediate allergic reaction or delayed skin reaction to an iodinated contrast material or any serious doubt about such a history.
* Pregnancy or breastfeeding in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Iohexol pharmacokinetic calculated with Bayesian estimator and with classic method | Hours: 0h30, 1h00, 1h30, 02h00, 03h00, 04h00, 05h00, 06h00, 09h00, 12h00 after Iohexol administration
  Clearance of Iohexol calculated with Bayesian estimator (limited samples) and with classic method (rich samples).

SECONDARY OUTCOMES:
Iohexol pharmacokinetic calculated with Bayesian estimator and Brochner-Mortensen method | Hours: 0h30, 1h00, 1h30, 02h00, 03h00, 04h00, 05h00, 06h00, 09h00, 12h00 after Iohexol administration
  Clearance of Iohexol calculated with Bayesian estimator (limited samples) and Brochner-Mortensen method (5 samples).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MARIAT, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No